CLINICAL TRIAL: NCT06386146
Title: A Phase 1/2a, Multi-Center, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-30355 in Adult Patients With Advanced Solid Tumors Harboring TP53 Y220C Mutation
Brief Title: JAB-30355 in Patients With Advanced Solid Tumors Harboring TP53 Y220C Mutation
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JAB-30355-1001
Record Dates: First submitted 2024-04-23; First posted 2024-04-26 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Solid Tumors
Keywords: TP53 Y220C reactivator; TP53 Y220C mutation; P53; Tumor protein p53; TP53; Advanced solid tumors; Ovarian Cancer; JAB-30355
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose escalation phase (Experimental): Multiple dose levels of JAB-30355 will be explored to determine the maximum tolerated dose (MTD)
  Interventions: Drug: JAB-30355
- Dose expansion phase (Experimental): Dose Expansion Phase will explore JAB-30355's clinical benefit and optimal tolerability in selected dose level.
  Interventions: Drug: JAB-30355

INTERVENTIONS:
Drug: JAB-30355 — Oral administration
  Arms: Dose escalation phase
Drug: JAB-30355 — Oral administration
  Arms: Dose expansion phase

SUMMARY:
This study is to evaluate the efficacy and safety of JAB-30355 in adult participants with advanced solid tumors harboring TP53 Y220C mutation.

DETAILED DESCRIPTION:
This study consists of two parts: Dose Escalation Phase (Phase 1) and Dose Expansion Phase (Phase 2a). The primary objective of dose escalation is to evaluate the safety and tolerability, and to determine the MTD of JAB-30355 monotherapy administered in participants with advanced solid tumors harboring TP53 Y220C mutation. Dose expansion will further explore JAB-30355's clinical benefit and tolerability in selected dose levels.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Participant must be ≥18 years of age at the time of signing the Informed Consent Form (ICF).
* ECOG performance status score of 0 or 1.
* Has been treated with at least one line of systemic therapy for that tumor type and stage.
* Have documentation of confirmed TP53 Y220C mutation.
* At least 1 measurable lesion per RECIST v1.1.
* Adequate hematological, renal and hepatic function and appropriate coagulation condition.
* Able to swallow and retain orally administered medication.

Exclusion Criteria:

* Active brain or spinal metastases or primary CNS tumor.
* Active infection requiring systemic treatment within 7 days.
* Active HBV or HCV.
* Any severe and/or uncontrolled medical conditions.
* LVEF ≤50% assessed by ECHO or MUGA.
* QTcF>470 msec.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2024-07-24 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Approximately one year
  Number and proportion of participants who experience at least one dose limiting toxicity (DLT)
Number of participants with adverse events | Approximately three years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms et al.

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) | Approximately three years
  Observed maximum plasma concentration after administration. Plasma concentrations of JAB-30355 from subjects will be used to calculate PK parameters.
Time to reach the observed maximum (peak) concentration (Tmax) | Approximately three years
  Time to reach the observed maximum (peak) concentration. Plasma concentrations of JAB-30355 from subjects will be used to calculate PK parameters.
Terminal half-life (t1/2) | Approximately three years
  Terminal half-life of JAB-30355 in human. Plasma concentrations of JAB-30355 from subjects will be used to calculate PK parameters.
Objective response rate (ORR) | Approximately three years
  ORR is defined as the percentage of participants with partial response (PR) or complete response (CR) based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of response (DOR) | Approximately three years
  DOR is defined as the time from the date of the first documented response (CR or PR) to the earliest date of disease progression or death, whichever occurs first, as determined by investigator assessment per RECIST v1.1.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (7):
  - Research Site, Denver, Colorado
  - Research site, Lake Mary, Florida
  - Research site, St Louis, Missouri
  - Research site, Canton, Ohio
  - Research site, Cleveland, Ohio
  - Research Site, Nashville, Tennessee
  - Research site, Houston, Texas
- China (4):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Jinan, Shandong
  - Research Site, Shanghai, Shanghai Municipality